CLINICAL TRIAL: NCT02955459
Title: VNRX-5133-101/102: A Randomized, Double Blind, Placebo-Controlled, Sequential Group, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Repeat Doses of VNRX-5133 in Healthy Adult Volunteers
Brief Title: VNRX-5133 SAD/MAD Safety and PK in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Venatorx Pharmaceuticals, Inc. (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: VNRX-5133-101/102; DMID 16-0014 (Other: DMID); 272201300019C-3-0-1 (NIH)
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Bacterial Infections
Keywords: Healthy volunteers; Pharmacokinetics
MeSH Terms: conditions — Bacterial Infections | interventions — taniborbactam

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- VNRX-5133 (Experimental): IV infusion
  Interventions: Drug: VNRX-5133
- Placebo (Placebo Comparator): IV infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VNRX-5133
  Arms: VNRX-5133
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a 2-part, first-in-human dose-ranging study to evaluate the safety, tolerability and pharmacokinetics of escalating doses of VNRX-5133 administered via intravenous (IV) infusion in healthy subjects. In part 1, subjects will receive a single dose of VNRX-5133; in part 2 subjects will receive VNRX-5133 for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Males or non-pregnant, non-lactating females
* Body Mass Index (BMI) between 18.5 - 32.0, inclusive.
* Suitable veins for cannulation

Exclusion Criteria:

* Employee of site or the sponsor
* Any disease that poses an unacceptable risk to participants
* Abnormal ECG
* Abnormal labs
* Abnormal vital signs
* Current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, autoimmune, hematologic, neoplastic, or neurological disorder
* Positive serology for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV) type 1
* Current smokers or history of smoking within 30 days

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2016-11; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events; assessed by patient reporting, physical exams, collection of vital signs, ECGs and absolute values and changes over time of hematology, chemistry and urinalysis. | Part 1: 8 days. Part 2: 17 days

CONTACTS AND LOCATIONS:
Locations (1):
- Lenexa, Kansas, United States

REFERENCES:
- [Derived] Dowell JA, Dickerson D, Henkel T. Safety and Pharmacokinetics in Human Volunteers of Taniborbactam (VNRX-5133), a Novel Intravenous beta-Lactamase Inhibitor. Antimicrob Agents Chemother. 2021 Oct 18;65(11):e0105321. doi: 10.1128/AAC.01053-21. Epub 2021 Aug 9. PMID 34370573